CLINICAL TRIAL: NCT02474680
Title: Evaluation of Pharmacogenetic Testing In a Mental Health Population and Economic Outcomes
Acronym: PGx-TIME
Status: Completed | Type: Observational
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: AIHG-1420-PGxTIME
Record Dates: First submitted 2015-02-05; First posted 2015-06-18 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Major Depressive Disorder 1
Keywords: depression; Major Depressive Disorder; MDD; mental health; pharmacogenomics; personalized medicine; precision medicine; anti-depressants
MeSH Terms: conditions — Major Depressive Disorder 1; Depression; Depressive Disorder, Major; Psychological Well-Being | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Care Coordination Group: Patients participating in the Avera Care Coordination Program for Intervention 'Pharmacogenetic testing'
  Interventions: Genetic: Pharmacogenetic testing

INTERVENTIONS:
Genetic: Pharmacogenetic testing — Psychotropic genotyping panel

SUMMARY:
This is a non-randomized, single-case design of pharmacogenetic implementation in a mental health patient population of subjects taking antipsychotics and/or antidepressants.

DETAILED DESCRIPTION:
This is a non-randomized, single-case design of pharmacogenetic implementation in a mental health patient population of subjects taking antipsychotics and/or antidepressants. Retrospective and prospective data will be collected on all subjects before and after pharmacogenetic recommendations have been made. Retrospective data will be collected for the previous 12 months before pharmacogenetic recommendations are made and prospective data will be collected for 12 months after pharmacogenomic recommendations have been made.

ELIGIBILITY:
Inclusion Criteria:

* Must be taking either an anti-depressant or an anti-psychotic medication
* Must provide informed consent
* Must have Avera Health Plans insurance coverage
* Must have three months of participation in the Avera Care Coordination Program

Exclusion Criteria:

* Must not be pregnant or breastfeeding
* Must not have an active and/or unstable diagnosis of substance abuse
* Must not have a primary diagnosis of dementia, bulimia, or anorexia nervosa disorder
* Must not have had a previous pharmacogenetic evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must be enrolled in the Avera Care Coordination Program and have insurance coverage through the Avera Health Plans
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Depression scores | 12 months
  Compare depression scores at baseline and following pharmacogenetic-guided medication recommendation

SECONDARY OUTCOMES:
Economic impact of pharmacogenetic testing | 12 months
  Data from patients' insurance provider will be compared pre- and post-pharmacogenetic testing. Such data may include hospitalizations, clinic visits, ER visits, medication expenses, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Stanely, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Institute for Human Genetics, Sioux Falls, South Dakota, United States